CLINICAL TRIAL: NCT04856098
Title: A Pharmacokinetic Feasibility Study on Ultibro Breezhaler, an Indacaterol-glycopyrronium Inhalation Powder Capsule, in Healthy Subjects
Brief Title: Absorption of Indacaterol and Glycopyrronium From Ultibro Breezhaler
Acronym: FINDA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 3131001
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Glycopyrrolate; Charcoal

STUDY DESIGN:
Intervention Model Description: The study is a 2-part crossover study where the study subjects participate either in part 1 (18 subjects) or in part 2 (16 subjects). The parts can run in sequence or in parallel. The study subjects in part 1 receive single doses of Ultibro Breezhaler on 3 periods and the study subjects in part 2 receive single doses of Ultibro Breezhaler on 2 periods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 Ultibro Breezhaler 2 capsules, Batch A (Experimental)
  Interventions: Drug: Indacaterol maleate and glycopyrronium bromide
- Part 1 Ultibro Breezhaler 2 capsules with charcoal, Batch A (Experimental)
  Interventions: Drug: Indacaterol maleate and glycopyrronium bromide; Drug: Ultibro Breezhaler with oral charcoal
- Part 1 Ultibro Breezhaler 1 capsule, Batch A (Experimental)
  Interventions: Drug: Indacaterol maleate and glycopyrronium bromide
- Part 2 Ultibro Breezhaler 2 capsules, Batch A (Experimental)
  Interventions: Drug: Indacaterol maleate and glycopyrronium bromide
- Part 2 Ultibro Breezhaler 2 capsules, Batch B (Experimental)
  Interventions: Drug: Indacaterol maleate and glycopyrronium bromide

INTERVENTIONS:
Drug: Indacaterol maleate and glycopyrronium bromide — Batch A Ultibro Breezhaler 85/43 μg 2 capsules
  Arms: Part 1 Ultibro Breezhaler 2 capsules with charcoal, Batch A; Part 1 Ultibro Breezhaler 2 capsules, Batch A; Part 2 Ultibro Breezhaler 2 capsules, Batch A
Drug: Indacaterol maleate and glycopyrronium bromide — Batch A Ultibro Breezhaler 85/43 μg 1 capsule
  Arms: Part 1 Ultibro Breezhaler 1 capsule, Batch A
Drug: Indacaterol maleate and glycopyrronium bromide — Batch B Ultibro Breezhaler 85/43 μg 2 capsules
  Arms: Part 2 Ultibro Breezhaler 2 capsules, Batch B
Drug: Ultibro Breezhaler with oral charcoal — Activated charcoal suspension, granules 50 g / bottle
  Arms: Part 1 Ultibro Breezhaler 2 capsules with charcoal, Batch A

SUMMARY:
The objective of this study is to assess pharmacokinetics (PK) of indacaterol and glycopyrronium, and methodology and practical arrangements for future studies.

ELIGIBILITY:
Main inclusion criteria:

1. Healthy males and females
2. 18-60 years of age
3. Body mass index 19-30 kg/m2
4. Weight at least 50 kg
5. Written informed consent obtained

Main exclusion criteria:

1. Evidence of a clinically significant cardiovascular, renal, hepatic, haematological, GI, pulmonary, metabolic, endocrine, neurological or psychiatric disease
2. Any condition requiring regular concomitant treatment
3. Any clinically significant abnormal laboratory value, vital sign or physical finding that in the opinion of the investigator could interfere with the interpretation of study results or cause a health risk for the subject
4. Known hypersensitivity to indacaterol or glycopyrronium
5. Pregnant or lactating females and females of childbearing potential not using contraception of acceptable effectiveness
6. Blood donation or loss of significant amount of blood within 90 days prior to the first study treatment administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Peak indacaterol concentration in plasma (Cmax) | between 0-72 hours after dosing
Peak glycopyrronium concentration in plasma (Cmax) | between 0-72 hours after dosing
Indacaterol area under the concentration-time curve from time zero to 30 minutes (AUC30min) | 0-30 minutes after dosing
Glycopyrronium area under the concentration-time curve from time zero to 30 minutes (AUC30min) | 0-30 minutes after dosing
Indacaterol area under the concentration-time curve from time zero to 72 hours (AUC72h) | 0-72 hours after dosing
Glycopyrronium area under the concentration-time curve from time zero to 72 hours (AUC72h) | 0-72 hours after dosing

SECONDARY OUTCOMES:
Indacaterol area under the concentration-time curve from time zero to the last sample with a quantifiable concentration (AUCt) | 0-18 days after dosing
Glycopyrronium area under the concentration-time curve from time zero to the last sample with a quantifiable concentration (AUCt) | 0-18 days after dosing
Indacaterol area under the concentration-time curve from time zero to infinity (AUCinf) | 0-18 days after dosing
Glycopyrronium area under the concentration-time curve from time zero to infinity (AUCinf) | 0-18 days after dosing
Time to reach peak indacaterol concentration in plasma | between 0-72 hours after dosing
Time to reach peak glycopyrronium concentration in plasma | between 0-72 hours after dosing
Indacaterol terminal elimination half-life (t1/2) | 0-18 days after dosing
Glycopyrronium terminal elimination half-life (t1/2) | 0-18 days after dosing
Number of adverse events as event counts and subjects counts | throughout the study, average 9-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Orion Corporation Clinical Study Director, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- CRST Helsinki Oy, Helsinki, Finland